CLINICAL TRIAL: NCT05213650
Title: Comparative Evaluation of Cleaning Agents on Color and Roughness of Invisalign Clear Aligners: A Cross-Over Randomized Trial
Brief Title: Cleaning Agents Impact on Invisalign Aligners: A Cross-Over Randomized Trial
Acronym: İnvisalign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Banu Kılıç, Assistant Professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BezmialemVU invisalign
Record Dates: First submitted 2022-01-17; First posted 2022-01-28 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Aligner Staining

STUDY DESIGN:
Intervention Model Description: controlled clinical trial
Who Masked: Participant
Masking Description: It will be shared with the participants of the study that when their treatment is finished, the plaques will be requested back and a study will be carried out on these plaques to affect the plaques from the process. However, the information that the study is on the effects of the cleaning agent they use will not be shared. Therefore, the participants do not have information about being in a group related to plaque cleaning efficiency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Invisalign control patients (liquid soap) (No Intervention): Patients who clean their plaques only with liquid soap and toothbrush
- Invisalign non-abrasive toothpaste patients (Experimental): Patients who clean their plaque with non-abrasive toothpaste and toothbrush
  Interventions: Other: non-abrasive toothpaste
- Invisalign abrasive toothpaste patients (Experimental): Patients who clean their plaque with abrasive toothpaste and toothbrush
  Interventions: Other: abrasive toothpaste
- Invisalign Efferdent patients (Experimental): Patients who clean their plaques with liquid soap and use Efferdent antibacterial cleaning tablet once a week
  Interventions: Other: Efferdent
- Invisalign Cleaning Crystals patients (Experimental): Patients who clean their plaques with liquid soap and use Invisalign Cleaning Crystals tablet once a week
  Interventions: Other: Cleaning Crystals

INTERVENTIONS:
Other: non-abrasive toothpaste — Aligners should be cleaned at least once a day, but twice is preferred to prevent them from changing color or having a bad odor. They should be treated just like teeth and cleaned often, especially after eating and drinking.Usually, dentists advise their patients to clean their plaques with only liquid soap, toothbrush and water. Non-abrasive toothpaste will be used as intervention to aligner cleaning during invisalign treatment.
  Other Names: cleaning agent
  Arms: Invisalign non-abrasive toothpaste patients
Other: abrasive toothpaste — Aligners should be cleaned at least once a day, but twice is preferred to prevent them from changing color or having a bad odor. They should be treated just like teeth and cleaned often, especially after eating and drinking.Usually, dentists advise their patients to clean their plaques with only liquid soap, toothbrush and water. Abrasive toothpaste will be used as intervention to aligner cleaning during invisalign treatment.
  Other Names: cleaning agent
  Arms: Invisalign abrasive toothpaste patients
Other: Efferdent — Aligners should be cleaned at least once a day, but twice is preferred to prevent them from changing color or having a bad odor. They should be treated just like teeth and cleaned often, especially after eating and drinking.Usually, dentists advise their patients to clean their plaques with only liquid soap, toothbrush and water.The Efferdent tablet will be used once a week as an intervention to aligner cleaning during invisalign treatment.
  Other Names: cleaning agent
  Arms: Invisalign Efferdent patients
Other: Cleaning Crystals — Aligners should be cleaned at least once a day, but twice is preferred to prevent them from changing color or having a bad odor. They should be treated just like teeth and cleaned often, especially after eating and drinking.Usually, dentists advise their patients to clean their plaques with only liquid soap, toothbrush and water. Invisalign Cleaning Crystals will be used once a week as an intervention to aligner cleaning during invisalign treatment.
  Other Names: cleaning agent
  Arms: Invisalign Cleaning Crystals patients

SUMMARY:
Today, the increasing aesthetic expectations of the patients, showing its effect in the field of orthodontics, leads to the orientation towards aesthetic materials. The Invisalign system is also polyurethane for aesthetic purposes.

It is a series of transparent plaques personalized to the patient's problems. However, the transparent structure of the plaque increases the importance of its cleanliness.

There are many studies evaluating the removal of bacterial biofilm from plaques. However There are minimal studies evaluating the effect of the materials used for cleaning on the light transmittance, which has a significant effect on the aesthetics of the plaques.

The aim of this study is to compare 5 different agents' effects on colour change.

The work created will be divided into 5 groups according to the cleaning materials used.

One of the cleaning agents will be assigned by lot and will be used while the treatment processes are continuing.

The colour measurement will be carried out using the VITA Easyshade Compact spectrophotometer (VITA Zahnfabrik DEASYC220, Bad Sackingen, Germany). To prevent external light interference and keep the measurement head in a fixed position for each measurement, a special cubic box with a 3 mm radius entrance was created. The head of the device was firmly attached to the box lid with black tape to increase light-tightness. The colour measurement will be performed from the occlusal region of the second premolar tooth on the aligners, which will be placed on a standard white background. The colour measurement will be carried out as received and after the aligners were used in the patient's mouth for 2 weeks. Prior to measurements, the spectrophotometer will be calibrated according to the manufacturer's instructions. Each measurement will be repeated three times, and the average value will be determined. The Commision de l'Eclairage (CIE) Lab* system will be used for colour measurements. This system uses three parameters to define colour. The L* coordinate is a brightness measure that ranges from 0 (black) to 100 (white); the a* coordinate is horizontal and shows chromatic coordinates between red (+) and green (-), and the b* coordinate is also horizontal and extends in the direction of yellow (b+) and blue (b-). To determine the colour difference, a formula (Formula 1) will be used. ∆L, ∆a, and ∆b values will be calculated by subtracting the starting measurements (L0, a0, b0) from the final measurements (L1, a1, b1). The ∆E value will be calculated using these values, and the colour difference between groups will be compared.

∆E2-1 = [(∆L)2 + (+ (∆a)2 + (∆b)2]1/2= [(L1-L0)2 + (a1-a0)2 + (b1-b0)2]1/2 The formula proposed by Filho and da Silva will be used to convert ΔE values to National Bureau of Standards (NBS) values. NBS unit = ΔE* × 0.92. The ΔE values will be converted to their clinical significance using the NBS system.

According to the results of the research, the colour change of the agents used to clean Invisalign aligners will be determined.

The use of agents that have a minor effect on aesthetics can be considered ideal according to the results of the study

DETAILED DESCRIPTION:
In recent years, following the developments in the field of orthodontics, the participation and expectations of patients in treatment have also changed. Conventional orthodontic brackets may cause aesthetic concerns in patients. The use of aesthetic materials and techniques aimed at overcoming such limitations has increased.

An orthodontic treatment system made with a material made of polyurethane was introduced for the first time in 1998 as an alternative to conventional brackets. This system uses CAD/CAM technology to produce serial plates personalized to the treatment process.

It is very important to clean these appliances for aesthetic reasons and to prevent bacteria from accumulating and becoming a focus of infection for the oral cavity. If plaques are not cleaned regularly, they can act as a reservoir for bacteria, leading to periodontal diseases, cavities and bad breath.

In the treatment of clear plaque, the patient is asked not to eat or drink anything other than water while the plaques are in the mouth. However, despite all the recommendations, patients sometimes do not comply with these and may consume coloring drinks while the plaques are in their mouths. This situation causes changes in the polymer of the material and adversely affects the aesthetics, which is the main advantage of clear aligner treatment.

Color stability of clear aligners remain critical considerations for both patients and clinicians. Despite the increasing cost, patients' desire for transparent aligners is due to the fact that these plates have almost no transparency in the mouth, so maintaining the original colour of the aligners is an important issue.

Although there are many studies in the literature evaluating the removal of bacterial biofilm after cleaning of clear plaques, there are very limited studies evaluating the Colour change of plaques.

In the light of this information, the aim of this research is to evaluate the colour change of transparent plaques, which is a polyurethane material, using 5 different cleaning methods. The cleaning methods to be used for this; toothpaste, whitening toothpaste, Corega Pro Guard & Retainer cleaning tablet, Efferdent antibacterial cleaning tablet and liquid soap.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study:

  1. No active periodontal disease
  2. No caries
  3. No systemic disease
  4. Patients who do not use any medication will be included in the study.
  5. Patients who will use more than 20 transparent plates in their treatment-

Exclusion Criteria:

1. Smoking (more than 1 pack per day)
2. Patients consuming dyes such as coffee, tea, beer and red wine more than 2 times a day
3. Patients using less than 20 clear plates in their treatment

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Colour change (Delta E)_control | 2 week
  Delta E of 12 clear aligners of patients who clean their plaques only with liquid soap and a toothbrush
Colour change (Delta E)_Invisalign non-abrasive toothpaste patients | 2 week
  Delta E of 12 clear aligners of patients who clean their plaques with non-abrasive toothpaste and toothbrush
Colour change (Delta E)_ Invisalign abrasive toothpaste patients | 2 week
  lDelta E of 12 clear aligners of patients who clean their plaque with abrasive toothpaste and toothbrush
Colour change (Delta E) Invisalign Efferdent patients | 2 week
  Delta E of 12 clear aligners of patients who clean their plaques with liquid soap and use Efferdent antibacterial cleaning tablet once a week
Colour change (Delta E) Invisalign Cleaning Crystals patients | 2 week
  Delta E of 12 clear aligners of patients who clean their plaques with liquid soap and use Invisalign Cleaning Crystals tablet once a week

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kılıç, Study Director — Bezmialem Vakıf Üniversitesi
Locations (1):
- Banu Kılıç, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papadimitriou A, Mousoulea S, Gkantidis N, Kloukos D. Clinical effectiveness of Invisalign(R) orthodontic treatment: a systematic review. Prog Orthod. 2018 Sep 28;19(1):37. doi: 10.1186/s40510-018-0235-z. PMID 30264270
- [Background] Kravitz ND, Kusnoto B, BeGole E, Obrez A, Agran B. How well does Invisalign work? A prospective clinical study evaluating the efficacy of tooth movement with Invisalign. Am J Orthod Dentofacial Orthop. 2009 Jan;135(1):27-35. doi: 10.1016/j.ajodo.2007.05.018. PMID 19121497
- [Derived] Kilic B, Canpolat S, Ozturk M. Comparative evaluation of the effect of different cleaning agents on colour and surface roughness of Invisalign clear aligners: a cross-over randomized controlled trial. BMC Oral Health. 2025 Nov 4;25(1):1745. doi: 10.1186/s12903-025-06928-w. PMID 41188779